CLINICAL TRIAL: NCT06633978
Title: A Pilot Study of the Impact of Personalized Digital Meditation on Improving Sleep and Reducing Stress in MCI
Brief Title: Studying the Effects of Digital Interventions on Cognition, Wellbeing, Stress, and Sleep in Older Adults
Acronym: MediDream
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AG083503; R61AG083503 (NIH)
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: MCI; Aging
Keywords: meditation; sleep; stress; attention; cognition; memory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- MediTrain (Experimental)
  Interventions: Device: MediTrain; Device: wrist worn multi-sensor watches; Device: Sleep monitor

INTERVENTIONS:
Device: MediTrain — Participants will engage with a digital meditation app for 30m/day for 6wks. MediTrain is a tablet-based, meditation-inspired, cognitive training game aimed at improving self-regulation of internal attention and distractions. It was developed in collaboration with meditation thought-leader Jack Kornfield, and Zynga, a world-class video game company. It was created to make benefits of concentrative meditation more easily accessible to anyone, including complete novices. This is achieved by creating a game that yields quantifiable and attainable goals, provides feedback, and includes an adaptive algorithm to gradually increase difficulty as users improve.
Device: wrist worn multi-sensor watches — Stress and sleep data will be recorded at home throughout the intervention using FDA-approved wrist worn multi-sensor watches.
Device: Sleep monitor — Sleep Profiler devices are FDA-cleared reduced-montage EEG recording devices that will be used in accordance with its FDA clearance. They are completely non-invasive and are designed to be comfortable enough to wear all night without interfering with normal sleep. These devices enable quality sleep recordings in the comfort of people's homes, rather than required an overnight stay at a sleep lab at UCSF.

SUMMARY:
The goal of this proposed research is to collect pilot data to test the hypothesis that treatment with a novel form of closed-loop digital meditation (MediTrain) will lead to a greater magnitude of gains in cognitive abilities in patients with mild cognitive impairment (MCI), compared to OA without cognitive impairment, and will lead to improvements in quantitative measures of sleep.

ELIGIBILITY:
comfortably ambulatory healthy physical condition normal or corrected to normal visual auditory acuity fluency in spoken English Between 60-85 years old No neurological or psychiatric disorders No substance abuse Not taking anti-depressants Not taking anti-anxiety medication No history of seizures No color blindness No glaucoma No macular degeneration No amblyopia (lazy eye) No strabismus (cross eyed) Aneurysm clip(s) No Cardiac pacemaker No Implanted cardioverter defibrillator (ICD) No Electronic implant or device No Magnetically-activated implant or device No Neurostimulation system No Spinal cord stimulator No Internal electrodes or wires No Bone growth/bone fusion stimulator No Cochlear, otologic, or other ear implant No Insulin or other infusion pump No Implanted drug infusion device No type of prosthesis (eye, penile, etc.) No Heart valve prosthesis No Eyelid spring or wire No Artificial or prosthetic limb No Metallic stent, filter, or coil No Shunt (spinal or intraventricular) No Vascular access port and/or catheter No Radiation seeds or implants No Swan-Ganz or thermodilution catheter No Medication patch (Nicotine, Nitroglycerine) No metallic fragment or metallic foreign body in/on the body that can not be removed No Wire mesh implant No Tissue expander (e.g., breast) No Surgical staples, clips, or metallic sutures No Joint replacement (hip, knee, etc.) No Bone/joint pin, screw, nail, wire, plate, etc. No IUD, diaphragm, or pessary No Dentures or partial plates that can not be removed No Tattoo or permanent makeup No Body piercing jewelry No Claustrophobia

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Mean change on the Continuous Performance Task (CPT) over time | baseline, immediate follow-up, and at a 6 month follow-up in a subset of participants
Mean change in sleep quality | baseline, immediate follow-up, and at a 6 month follow-up in a subset of participants
  Mean change in sleep quality (i.e., total sleep time / time in bed, therefore this measure incorporates latency to sleep onset, total sleep time, wake after sleep onset and early morning waking, with higher numbers associated with better sleep) over time [Time Frame: baseline, immediate follow-up, and at a 6 month follow-up in a subset of participants]
Mean change in measures of stress reactivity over time | baseline, immediate follow-up, and at a 6 month follow-up in a subset of participants
  Measures of heart rate variability (HRV) and electrodermal activity (EDA) while participants perform a stress-inducing task

SECONDARY OUTCOMES:
Mean change in Telomere length (quantified in peripheral blood cells) over time | baseline, immediate follow-up, and at a 6 month follow-up in a subset of participants
  200 mL of blood will be collected from each participant before and after the intervention. Blood will be centrifuged for whole blood cell acquisition and stored at -80 °C for subsequent batch testing. Telomere length (T/S ratio) will be quantified in peripheral blood mononuclear cells.
Mean change on a distracted attention task over time | baseline, immediate follow-up, and at a 6 month follow-up in a subset of participants
  Mean performance on a distracted attention task will be compared pre and post intervention. Divided attention performance will be assessed using the Filter Task that places simultaneous demands on perceptual discrimination abilities and distraction filtering.
Mean change in Frontal Theta Power over time | baseline, immediate follow-up, and at a 6 month follow-up in a subset of participants
  Based on previous studies of meditation training and our preliminary data, we predict that MediTrain will lead to significantly enhanced midline frontal theta power during the TOVA in MCI as compared to OA. Beyond most prior studies, by collecting structural MRI data, we will be able to source-localize any observed changes in midline frontal theta.
Mean change in resting state networks over time | baseline, immediate follow-up, and at a 6 month follow-up in a subset of participants
  We also expect MediTrain will augment intrinsic Default Mode Network (DMN) connectivity, both functionally (measured with resting fMRI111,112) and structurally (measured with DTI-based connectomes). This is hypothesized based on the known association between the DMN,

OTHER OUTCOMES:
Mean change on the Adaptive Cognitive Evaluation (ACE) over time | baseline, immediate follow-up, and at a 6 month follow-up in a subset of participants
  The ACE is a mobile cognitive assessment tool, which includes a battery of cognitive control tests for rapid tests of cognition. The sub-tests (or 'modules') in ACE are adapted from standardized tasks to rapidly assess various aspects of cognition, including attention, memory, and multitasking. We will assess response time, accuracy, and response time variability in each case, with faster/more accurate/less variable performance being indicative of improved cognitive control, meditation, and frontal theta power.
Mean change in continuous recordings of sleep metrics. | baseline, immediate follow-up, and at a 6 month follow-up in a subset of participants
  We will assess time spent in NonREM stages 1 (N1), 2 (N2) and 3 (N3) sleep and REM sleep (RS), latency to sleep onset (SOL), and wake after sleep onset (WASO). We will also assess delta power during sleep stages and wake; and overall sleep maintenance (SM) and sleep efficiency (SE). Diminished time spent in SOL and WASO, increased time N2, N3 and REM sleep, increased delta during NonREM sleep are each signs of improved sleep. Increases in SM and SE indicated improved, more stable sleep patterns
mean change in Change in Mnemonic Discrimination over time | baseline, immediate follow-up, and at a 6 month follow-up in a subset of participants
  Mnemonic discrimination task tests recognition memory for common objects, as reported in scores on a scale of the Lure Discrimination Index ranging from 0.00 to 1.00 where higher values show better performance.
mean change in Task-based Cortical Functional Connectivity | baseline, immediate follow-up, and at a 6 month follow-up in a subset of participants
  functional MRI data associated With Training-induced Changes in Mnemonic Discrimination will be analyzed in terms of beta-series correlations between co-active cortical regions of interest and compared between treatment arms and timepoints.
Mean Change on Everyday Cognition Scale (ECog) | baseline, immediate follow-up, and at a 6 month follow-up in a subset of participants
  The Everyday Cognition Scale (ECog) measures the ability to perform everyday tasks that demand memory, language, visuospatial abilities, planning, organization, and divided attention. The ECog consists of a global and domain scores for each of the previously described categories, and is scored as follows: 1= better or no change compared to 10 years earlier, 2= questionable/occasionally worse compared to 10 years earlier, 3= consistently a little worse compared to 10 years earlier, 4= consistently much worse compared to 10 years earlier. Thus, the lower the overall score is on this measure at both the global and domain score level, the better one is performing with respect to their cognition.
Mean Change on SF-36 (overall health) | baseline, immediate follow-up, and at a 6 month follow-up in a subset of participants
  SF-36 (overall health) The general health and well-being (SF-36) score assesses participant health. The SF-36 score ranges from 0 to 100. The higher the overall score is on this measure, the better one is performing with respect to their health and well-being.
Mean Change on Perceived Stress Scale | baseline, immediate follow-up, and at a 6 month follow-up in a subset of participants
  Perceived Stress Scale A survey that measures the degree to which situations in one's life are perceived as stressful. Scores range from 0 to 40 with higher scores representing more perceived stress. We will report change in means over time.
Mean Change on Pittsburgh Sleep Quality Index | baseline, immediate follow-up, and at a 6 month follow-up in a subset of participants
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete. Overall scores range from 0 to 21, with lower scores representing healthier sleep quality. We will report change in means over time.
Mean Change on Epworth Sleepiness Scale | baseline, immediate follow-up, and at a 6 month follow-up in a subset of participants
  The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life.
Mean Change on Profile of Mood States | baseline, immediate follow-up, and at a 6 month follow-up in a subset of participants
  POMS is a 65 questions psychometric instrument that measures the mood states of tension, depression, anger, vigor, fatigue, and confusion.
Mean Change on Berlin Questionnaire | baseline, immediate follow-up, and at a 6 month follow-up in a subset of participants
  The Berlin Questionnaire consists of 3 categories of questions related to the risk of having sleep apnea. Patients can be classified into High Risk or Low Risk based on their responses to the individual items and their overall scores in the symptom categories.
Mean Change on Insomnia Severity Index | baseline, immediate follow-up, and at a 6 month follow-up in a subset of participants
  The Insomnia Severity Index (ISI) is a brief screening tool for insomnia. It consists of seven questions regarding the nature and symptoms of sleep problems that respondents rate using a Likert scale ranging from 0 to 4. A total score of 0-7 indicates "no clinically significant insomnia," 8-14 means "subthreshold insomnia," 15-21 is "clinical insomnia (moderate severity)," and 22-28 means "clinical insomnia (severe).

CONTACTS AND LOCATIONS:
Overall Officials: David Ziegler, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No